CLINICAL TRIAL: NCT05085288
Title: The PROTECT 2 Study: Pressure Injury Treatment by Intermittent Electrical Stimulation: A Randomized, Controlled Trial
Brief Title: The PROTECT 2 Study : Pressure Injury Treatment by Intermittent Electrical Stimulation: A Randomized, Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21-1009
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2024-12

CONDITIONS: Stage 1 Pressure Ulcer; Stage 2 Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intermittent electrical stimulation system (IES) treatment Group (Active Comparator): Charged pulses will be administered to bilateral gluteus maximus through surface electrodes. Stimulation occurs at 30 Hz for 10 seconds every 10 minutes.
  Interventions: Device: Intermittent electrical stimulation system (IES) treatment and turning patient every two hours
- Standard of care Group (Active Comparator): Standard inpatient nursing practice for wound care, wound care prevention, and any other wound care or plastic surgery treatments deemed appropriate as per usual care.
  Interventions: Other: Turning population every two hours

INTERVENTIONS:
Device: Intermittent electrical stimulation system (IES) treatment and turning patient every two hours — The investigators propose to assess whether addition of the IES system and the use of standard of care wound care and wound prevention reduces the morbidity of sacral and ischial pressure injuries by decreasing progression of stage 1 and stage 2 ulcers or facilitates their healing compared to standard wound care in an inpatient critical care population.
  Arms: Intermittent electrical stimulation system (IES) treatment Group
Other: Turning population every two hours — The investigators propose to assess whether current standard of care wound care and wound prevention reduces the morbidity of sacral and ischial pressure injuries.
  Arms: Standard of care Group

SUMMARY:
Multicentered randomized controlled study with adaptive design to evaluate if Intermittent Electrical Stimulation (IES) decreases progression and facilitates healing of pressure injuries for patients with, sacral / ischial pressure injuries.

DETAILED DESCRIPTION:
This is a two-arm, prospective randomized control trial assessing whether IES combined with the standard of care (treatment) is superior to the standard of care alone (control). The study is a parallel design, adaptive, non-blinded randomized controlled trial, and uses two-sided analysis. We plan interim analyses at each 25% of the N. Part of the early interim analyses (first and second) will involve reassessing the a priori assumptions on data distributions and variability use in sample size calculations and updating the study size needed. Treatment effect results will be shared with the Data Safety Monitoring Board (DSMB) to determine whether the study should be ended early for either futility or having demonstrated superiority of the intervention. Patients can be entered into the protocol multiple times with independent assessments of inclusion/exclusion criteria and new consent for each enrollment. At each enrollment they will be re-randomized to either experimental or control arm. For the purpose of overall survival analysis (the only endpoint with a delayed assessment of outcome), such patients will be excluded.

This trial studies adult inpatients in both ICU and non-ICU environments with either new or established stage 1 or stage 2 sacral and ischial pressure injuries. Patients with a pacemaker/AICD, rhabdomyolysis, gluteal skin breakdown, and unstable fractures at risk of displacement by IES are excluded. Patients with atrial or ventricular wires after cardiac surgery can be enrolled as long as they are not being paced or in the opinion of the treating physician are at high risk of requiring pacing.

Subjects will be assessed for pressure injury status from point of randomization to discharge, death, or a minimum of 30 days. Device utilization and data collection can stop after 14 days in a non-ICU environment or when a total of 30 days of data collection has been met. If subjects are in the ICU longer than 30 days or when the combined total of ICU and less than 14 non-ICU days is greater than 30 days, the assessment and use of the device may continue after 30 days. Following entry into the study, participants will receive either the IES device in addition to the standard of care (treatment group) or the standard of care alone (control group). The study is expected to complete accrual within 12-18 months. Participant treatment will occur for the same amount of time as pressure injury assessment occurs as described above.

ELIGIBILITY:
Inclusion Criteria:

* Either new or established stage 1 or 2 sacral or ischial pressure ulcer in the ICU or non-ICU environments.
* Participants capable of giving informed consent, or if propitiate, participants having an acceptable individual capable of giving consent on the participant's behalf.

Exclusion Criteria:

* Unstable spinal, pelvic, or hip fractures that may be displaced by a forced contraction.
* Rhabdomyolysis
* Presence of permanent pacemaker or AICD, and for those with external wires after cardiac surgery, those who are using or at high risk for the development of a requirement for an external pacemaker.
* Skin breakdown or malignant skin involvement over the gluteal regions that would preclude the use of surface electrodes
* BMI > 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of adding the IES System to standard of care | 24 hours of admission to the ICU or non-ICU hospital service
  Investigators will assess the IES System to determine the efficacy of an IES system after being added to the standard of care on the primary outcome of sacral and ischial pressure injury score measured over time.
Compare using the IES oppose to only standard care | 24 hours of admission to the ICU or non-ICU hospital service
  Investigators will assess time to resolution of the ulcer

SECONDARY OUTCOMES:
Compare IES to standard care | 24 hours of admission to the ICU or non-ICU hospital service
  Time to resolution of ulcer
Evaluate treatment effect heterogeneity across levels of the following patient factors | 24 hours of admission to the ICU or non-ICU hospital service until discharged
  A variety of patient factors will be evaluated for treatment effect heterogeneity

CONTACTS AND LOCATIONS:
Overall Officials: Chase Donaldson, MD, Principal Investigator — The Cleveland Clinic; Andrea Kurz, MD, Study Chair — The Cleveland Clinic
Locations (3):
- United States (2):
  - Wake Forest Unverisity, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
- Univeristy of Graz, Graz, Austria

REFERENCES:
- [Derived] Donaldson C, de Abreu MG, Mascha EJ, Rowbottom J, Harvester E, Khanna A, Sura T, Sessler DI, Patarroyo FR, Gulluoglu A, Zajic P, Chauhan U, Essber H, Kurz A. Pressure injury treatment by intermittent electrical stimulation (PROTECT-2): protocol for a multicenter randomized clinical trial. Trials. 2024 May 10;25(1):313. doi: 10.1186/s13063-024-08085-x. PMID 38730383